CLINICAL TRIAL: NCT06817824
Title: The Effect of Su-Jok Therapy Applied to the Elderly on Constipation Symptoms and Quality of Life
Acronym: Su-Jok Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Leyla SEZGİN, Lecturer, Muş Alparslan University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: E-35465298-605-233507607
Record Dates: First submitted 2025-01-06; First posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Elderly (people Aged 65 or More); Quality of Life; Constipation
Keywords: elderly; constipation; sujok therapy
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: It is aimed to measure how it affects the quality of life as well as the improvement of constipation symptoms in the elderly after the application of Su Jok therapy. When the targeted data is reached, it is thought that it will contribute to the use of Su Jok therapy as a non-pharmacological method in the treatment of constipation in our country. In addition, since we are an aging country, the targeted group of individuals over the age of 65 is of particular importance. Since the population of the elderly is increasing, it is thought that the determination and application of alternative approaches that have a positive contribution to health and economic alternative approaches to improve the quality of life of the elderly will make significant contributions to both individuals and the ccountry's economy.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Over 65 years of age with constipation
- experiment (Experimental): Over 65 years of age with constipation
  Interventions: Other: Su-jok therapy

INTERVENTIONS:
Other: Su-jok therapy — Su Jok therapy was developed by South Korean scientist Professor Woo Jae Woo (1942-2010) in 1986. In Korean language, 'Su' means hand and 'Jok' means foot (Friman & Chelala, 2016; Ivanov 2018; Woo 1987, 1991, 2000, 2002, 2007; Sharma & Sharma, 2015). In Su Jok therapy, it is argued that there are reflection points of the body in the hands and feet and that these points activate every organ and part of the body like a remote control (Woo 1987, 1991, 2000, 2002, 2007; Şimşek & Alpar, 2020).
  Holistic approaches, energy flow and meridians form the basis of Su Jok therapy (Ivanov, 2018; Seth, 2013). Su Jok is an integrated therapy method that includes many tried and trusted methods of oriental medicine (Ponni, 2011; Rodríguez et al., 2018; Seth, 2013). In particular, it is similar in content to practices such as acupuncture and acupressure, which are approaches expressed by the same philosophy (Ivanov 2018; Ponni, 2011; Rodríguez et al., 2018).
  Arms: experiment

SUMMARY:
This article discusses the prevalence and health implications of constipation in the elderly population. Health problems increase with age and negatively affect quality of life. Constipation is a common problem in the elderly that severely reduces quality of life and is associated with many factors. Pharmacologic and non-pharmacologic methods are used for the management of constipation, but long-term use of pharmacologic treatments may lead to adverse effects. Therefore, non-pharmacologic approaches are gaining more importance.

In this context, Su Jok therapy, as an oriental medicine method, is a treatment method that aims to affect various organs of the body by using reflection points on the hands and feet. It is argued that Su Jok therapy can be beneficial in terms of symptom management and improving quality of life, especially in fields such as nursing and midwifery. In Turkey, there are no studies examining the effect of Su Jok therapy on constipation symptoms. This project aims to determine the effect of Su Jok therapy on constipation symptoms and quality of life, and the results are expected to contribute to the development of health services and treatment methods

DETAILED DESCRIPTION:
With the increase in chronic diseases in the elderly population, millions of people need nursing home and home care. Changes in health status with advancing age negatively affect the quality of life of the elderly and the elderly face many complex health problems. One of the common problems in the elderly is constipation. Diet low in fiber or fluids, immobility, general pain or discomfort, local pain due to hemorrhoids or anal fissure, medical problems such as irritable bowel syndrome or Parkinson's disease, drug treatments such as analgesics, antidepressants, psychiatric disorders such as depression, stress and changes in the individual's life cause constipation. Constipation is defined as infrequent defecation or difficulty in emptying the stool. It is associated with various symptoms such as hard stools, straining, feeling of anorectal obstruction, feeling of inadequate emptying, prolonged defecation time, unsuccessful defecation attempts, abdominal pain and bloating.

In addition to serious health problems, constipation has a serious negative impact on the quality of life of individuals that cannot be ignored. It is important to monitor and treat constipation, which is an important health problem in the elderly because it decreases the quality of life, causes loss of energy, increases health care costs and leads to serious medical problems. Therefore, it is extremely important to monitor constipation, to raise awareness about constipation in elderly individuals and to provide rapid treatment of constipation. Currently, pharmacologic and non-pharmacologic approaches are used in the management of constipation. In addition to medication (laxatives, suppositories, enemas), interventions such as biofeedback, acupressure, education, bowel habituation, exercise, yoga, aromatherapy, stress management and abdominal massage are generally utilized. Although the use of common pharmacological approaches in the management of constipation is effective in alleviating symptoms in the short term, long-term use of these agents may cause adverse effects such as diarrhea and metabolic disorders.

In addition, the fact that laxatives are costly and cause fluid, acid-base imbalance and electrolyte loss as a result of inappropriate use makes non-pharmacological methods necessary.

Su Jok therapy was developed by South Korean scientist Professor Woo Jae Woo (1942-2010) in 1986. In Korean, "Su" means hand and "Jok" means foot . In Su Jok therapy, it is argued that there are reflection points of the body in the hands and feet and that these points activate every organ and part of the body like a remote control.

Holistic approaches, energy flow and meridians form the basis of Su Jok therapy . Su Jok is an integrated therapy method that includes many tried and trusted methods of oriental medicine. In particular, it is similar in content to practices such as acupuncture and acupressure, which are approaches expressed by the same philosophy.

In the literature, it is argued that nurses can apply Su Jok therapy as an integrative method in symptom management for reasons such as the simplicity of the application of Su Jok therapy, which is similar to the philosophy of integrative nursing, the absence of any side effects and the absence of an interventional intervention. In our country, no study examining the effect of Su Jok Therapy on constipation symptoms has been found. In the study to be conducted within the scope of this project, it is aimed to determine the effect of Su Jok therapy on constipation symptoms and quality of life and to pioneer future research. The results obtained in the study in this project are thought to contribute significantly to the development of midwifery and nursing practices. When the data targeted in the study are reached, it is aimed to use Su Jok therapy as a non-pharmacological method in our country, and also to improve constipation symptoms and quality of life in preventive, curative and therapeutic health service provision.

ELIGIBILITY:
Inclusion Criteria:

* Young individuals aged 65-74 years, middle-aged individuals aged 75-84 years and hospitalised individuals aged 85 years and over who agreed to participate in the study,
* Scores of 24 and above on the Mini Mental Test,
* Those who score 3 points and above on the Visual Comparison Scale,
* Those who meet the Rome IV Criteria,
* Elderly people aged 65 years and over who do not have any lesion, infection, etc. that would prevent the application of Su Jok treatment on the hands and feet, who do not have acute diarrhoea, who do not have significant intestinal pathology such as incontinence and faecal impaction, who do not have inflammatory bowel disease, who have not had bowel surgery before, who do not use laxatives during the application will be included in the study.

Exclusion Criteria:

* Those who do not fulfil the inclusion criteria,
* Patients with cognitive impairment such as dementia and Alzheimer's,
* Patients with hearing problems or using hearing aids,
* Older people who did not want to participate in the study.

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2025-10-20 (Estimated); Study Completion 2025-10-20 (Estimated)

PRIMARY OUTCOMES:
The Effect of Su-Jok Therapy Applied to the Elderly on Constipation Symptoms | Regression of constipation symptoms in 3 months
  Rome IV Criteria Rome IV criteria are frequently used to diagnose functional constipation without an organic aetiology. Symptom-based Rome criteria were developed by an international team in line with the consensus of experts in the field . In the mid-1980s, more than 20 criteria were developed and a series of committee decisions were published by the Rome Committees convened to categorise and classify functional gastrointestinal disorders. These documents were subsequently updated and published as Rome I criteria in 1994. These criteria have been updated several times until today, and after 10 years of use of Rome III, the latest version of the criteria was published as Rome IV in May 2016 . Rome IV criteria are the most frequently used consensus definitions for clinical and research in the definition of constipation and can be easily understood and answered by patients.

SECONDARY OUTCOMES:
The Effect of Water Jok Therapy Applied to the Elderly on Quality of Life | Regression of constipation symptoms in 3 months
  Constipation Quality of Life Scale (QoLQS) It is the only scale originally developed to measure quality of life in individuals with constipation. Developed by Marquis et al. in 2005, the QoLQS has a total of 4 sub-dimensions and 28 questions, including 11 questions in the 'worry/anxiety' sub-dimension, 4 questions in the 'physical discomfort' sub-dimension, 8 questions in the 'psychosocial discomfort' sub-dimension, and 5 questions in the 'satisfaction' sub-dimension. Questions 18, 25, 26, 27 and 28 in the scale are calculated by reversing them. Scores that can be obtained from the 5-point Likert-type scale are between 28-140. The increase in the scores that can be obtained from the scale indicates that the quality of life is deteriorating.